CLINICAL TRIAL: NCT00120445
Title: Comparison of Air and Expansile Gas in Pneumatic Retinopexy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Yosanan Yospaiboon, Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE470116; TRF470116 (Other Grant/Funding Number: Thailand Research Fund)
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Retinal Detachment
Keywords: retinal detachment; pneumatic retinopexy
MeSH Terms: conditions — Retinal Detachment | interventions — Air

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Active Comparator): air vs perfluoropropane gas in pneumatic retinopexy
  Interventions: Procedure: air; Procedure: expansile gas

INTERVENTIONS:
Procedure: air — 0.3 ml of filtered air
Procedure: expansile gas — 0.3 ml of perfluoropropane gas

SUMMARY:
The objective of the study is to evaluate the results of using air versus expansile gas (perfluoropropane) in the treatment of rhegmatogenous retinal detachment by pneumatic retinopexy, comparing the retinal reattachment rate and post-operative visual recovery.

DETAILED DESCRIPTION:
To the best of the investigators' knowledge there have been no clinical trials to compare air and expansile gas in pneumatic retinopexy. The investigators hypothesize that both air and expansile gas have the same properties of gas and remain in the eye for 5-6 days which is long enough to have moderate chorioretinal adhesion to seal the retinal break. If the investigators can prove that air is equivalent to expansile gas in this procedure, it can save a lot of money for the country. Therefore, the investigators are conducting a randomised controlled double-blind study to compare the results of using air and perfluoropropane in pneumatic retinopexy for treatment of rhegmatogenous retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* Superior retinal break from 8 o'clock to 4 o'clock
* Single retinal break not greater than 2.5 clock hours in size
* Multiple breaks not greater than 3 clock hours away
* No (or minimal) proliferative vitreoretinopathy
* Physically and mentally co-operated in post-operative head positioning
* Signed informed consent form for the study

Exclusion Criteria:

* Ocular media opacities
* Advanced glaucoma
* Aphakia or pseudophakia
* Previous ocular surgeries
* One-eyed patients
* Subject did not sign informed consent form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2004-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
The retinal reattachment rate (calculated from the number of patients who had post-operative attached retinas divided by the total number of patients treated) | 1 week

SECONDARY OUTCOMES:
The final visual recovery (calculated from the difference between pre-operative and post-operative visual acuity) | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yosanan Yospaiboon, M.D., Principal Investigator — Khon Kaen University
Locations (1):
- Eye outpatients department, Srinagarind Hospital, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Result] Sinawat S, Ratanapakorn T, Sanguansak T, Prompol S, Laopaiboon M, Yospaiboon Y. Air vs perfluoropropane gas in pneumatic retinopexy: a randomized noninferiority trial. Arch Ophthalmol. 2010 Oct;128(10):1243-7. doi: 10.1001/archophthalmol.2010.230. PMID 20937993
- [Derived] Schwartz SG, Flynn HW Jr, Wang X, Kuriyan AE, Abariga SA, Lee WH. Tamponade in surgery for retinal detachment associated with proliferative vitreoretinopathy. Cochrane Database Syst Rev. 2020 May 13;5(5):CD006126. doi: 10.1002/14651858.CD006126.pub4. PMID 32408387